CLINICAL TRIAL: NCT01823653
Title: A Study to Investigate the Safety and Efficacy of Treatment of Subcutaneous Adipose Tissue in the Thighs Using the Liposonix System (Model 2)
Brief Title: Treatment of Subcutaneous Adipose Tissue in the Thighs Using High Intensity Focused Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solta Medical (Industry)
Responsible Party: Sponsor
Organization: Valeant Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-130-LP-H
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Treatment of Adipose Tissue in the Thighs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated Thigh (Experimental): Subjects randomly received treatment of either the left or right thigh with the Liposonix System (Model 2)
  Interventions: Device: Liposonix System (Model 2)

INTERVENTIONS:
Device: Liposonix System (Model 2) — Treatment of Subcutaneous Adipose Tissue in the thighs using High Intensity Focused Ultrasound

SUMMARY:
The purpose of this study is to assess the safety and efficacy of treatment with the Liposonix System (Model 2) for the circumferential reduction of subcutaneous adipose tissue (SAT) of the thighs.

DETAILED DESCRIPTION:
Subjects received a single treatment (Liposonix System) on one randomly assigned thigh. The opposite thigh was not treated and served as a control for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18-60 years of age
* Body Mass Index of ≤30 lb/in2
* Thickness of adipose tissue is at least 1.0 cm beyond the selected focal depth in the area to be treated (≥2.3cm)
* Subjects must agree not to alter their regular diet or exercise routines during the course of the study
* Subjects must be willing and able to comply with all study visit requirements, procedures, and assessments
* Subject must understand the nature of the study and sign an IRB approved Informed Consent

Exclusion Criteria:

* Subjects is pregnant
* Subjects diagnosed with a coagulation disorder or receiving anticoagulant therapy
* Subject has had prior aesthetic procedures in the area to be treated
* Subjects has pacemaker, defibrillator, or other implantable electrical device
* Subject has significant circumferential asymmetry between thighs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Van Dyke Laser and Skin, Paradise Valley, Arizona
  - Solta Medical Aesthetic Center, Hayward, California
  - Jewell Plastic Surgery Center, Eugene, Oregon
- Solish M.D., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Thigh: Randomly chosen left or right thigh treated with the Liposonix System (Model 2)
Period: Overall Study
Arm/Group | Treated Thigh
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Cohort
Arm/Group | Treated Thigh
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 58
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement in Thigh Circumference
Description: Clinical improvement measured by change from baseline thigh circumference after treatment
Time Frame: 12 weeks (minus baseline)
Population: Per Protocol
Measure: Least Squares Mean (Standard Error); unit: centimeter
Groups:
- Treated Thigh: Randomly assigned left or right thigh that received treatment with Liposonix System (Model 2)
- Control Thigh: Each subject's own thigh untreated during study
Arm/Group | Treated Thigh | Control Thigh
Number analyzed (Participants) | 58 | 58
centimeter | -1.22 (0.17) | -0.59 (0.17)

2. Secondary Outcome: Percentage of Participants Showing Clinical Improvement Using the Global Aesthetic Improvement Scale (GAIS) Post Treatment, Assessed by Investigator
Description: Investigator improvement at 12 weeks using the GAIS Scale, as presented based on percentage of subjects showing improvement. Outcome presented in % of participants that had GAIS scores of either 4 (improved) or 5 (much improved) at 12 weeks post treatment.
  *GAIS Scale: 1=Much Worse, 2=Worse, 3=No Improvement, 4=Improved, 5=Much Improved
Time Frame: 12 weeks
Population: Per protocol
Measure: Number; unit: Percentage of subjects improved
Arm/Group | Treated Thigh
Number analyzed (Participants) | 58
Percentage of subjects improved | 79.3

3. Secondary Outcome: Patient Satisfaction Using 1-5 Likert Scale
Description: Likert scale ranges from 1=Very Dissatisfied to 4=satisfied, 5=very satisfied. Percentage of participants rated 4 and 5 are reported below
Time Frame: 12 weeks
Population: Per protocol
Measure: Number; unit: percentage of subjects satisfied
Arm/Group | Treated Thigh
Number analyzed (Participants) | 58
percentage of subjects satisfied | 56.9

4. Secondary Outcome: Safety Assessment
Description: Discomfort level during treatment using the Visual Analog Scale (VAS) and post-treatment skin reponses or side effects using a 0-3 severity scale.
Time Frame: 1, 4, 8, 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Subcutaneous Adipose Thickness
Description: Ultrasound assisted measurement of adipose tissue thickness
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Score Post Treatment Assessed by Investigator for Determining Clinical Improvement
Description: Mean Investigator improvement at 12 weeks using the GAIS Scale.
  *GAIS Scale: 1=Much Worse, 2=Worse, 3=No Improvement, 4=Improved, 5=Much Improved
Time Frame: 12 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treated Thigh
Number analyzed (Participants) | 58
units on a scale | 3.8 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day 0 through study exit (12-weeks post treatment)
Arm/Group | Treated Thigh
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 26/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Thigh (N=60)
Ecchymosis (Skin and subcutaneous tissue disorders) | 7
Tenderness (Skin and subcutaneous tissue disorders) | 18
Dysesthesia (Skin and subcutaneous tissue disorders) | 3
Itchiness (Skin and subcutaneous tissue disorders) | 3
Discoloration (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall notify Sponsor of the intent to publish or present independent Study Data, and agrees not to publish or publicly present and/or discuss such data, Investigator's current findings and/or the results of the Study independently without the express written consent of Sponsor, which consent may be withheld. Sponsor reserves the right to require Investigator to remove any/all confidential information from any/all publications.